CLINICAL TRIAL: NCT01563601
Title: A Randomized, Open-Label Study to Evaluate the Efficacy and Safety of Obatoclax Mesylate in Combination With Carboplatin and Etoposide Compared With Carboplatin and Etoposide Alone in Chemotherapy-Naive Patients With Extensive-Stage Small Cell Lung Cancer
Brief Title: Efficacy and Safety of Obatoclax Mesylate in Combination With Carboplatin and Etoposide Compared With Carboplatin and Etoposide Alone in Chemotherapy-Naive Patients With Extensive-Stage Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C41601/3099; 2011-005591-41 (EudraCT Number)
Record Dates: First submitted 2012-03-15; First posted 2012-03-27 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Extensive-stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — obatoclax; Carboplatin; Etoposide; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Obatoclax mesylate, Carboplatin and Etoposide (CEO) (Experimental)
  Interventions: Drug: Obatoclax Mesylate, Carboplatine and Etoposide
- Carboplatin and Etoposide (CE) (Active Comparator)
  Interventions: Drug: Carboplatin and Etoposide

INTERVENTIONS:
Drug: Obatoclax Mesylate, Carboplatine and Etoposide — Obatoclax Mesylate:
  30 mg fixed dose;administered IV on days 1-3 every 21 days for 6 cycles. Maintenance therapy (optional and only if documented CR or PR) with obatoclax mesylate is administered at the same IV dose on days 1-3 every 21 days until disease progression or death.
  Carboplatin:
  Dose targeted at AUC of 5; administered IV on Day 1 only every 21 days for 6 cycles
  Etoposide:
  100mg/m2 administered IV on Days 1-3 every 21days for 6 cycles
  Other Names: Obatoclax: CEP-41601; Carboplatin: Paraplatin; Etoposide: Eposin, Neoposid, Vepesid, Etopophos
  Arms: Obatoclax mesylate, Carboplatin and Etoposide (CEO)
Drug: Carboplatin and Etoposide — Carboplatin:
  Dose targeted at AUC of 5 administered IV on Day 1 only every 21 days for 6 cycles.
  Etoposide:
  100mg/m2 administered IV on Days 1-3 every 21 days for 6 cycles
  Other Names: Carboplatin: Paraplatin; Etoposide: Eposin, Neoposid, Vepesid, Etopophos
  Arms: Carboplatin and Etoposide (CE)

SUMMARY:
This is a randomized, multi-center, open-label study of approximately 24 months duration (including follow up survival) to evaluate the safety and efficacy of obatoclax mesylate in combination with carboplatin and etoposide versus carboplatin and etoposide alone in chemotherapy-naive patients with extensive-stage small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patient has histologic or cytologic confirmation (upon local review) of small cell lung cancer (SCLC).
* The patient has extensive-stage small cell lung cancer (ES-SCLC), as defined by National Comprehensive Cancer Network (NCCN) guidelines.
* The patient has measurable disease as assessed by Response Evaluation Criteria Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1).
* The patient has not received any prior chemotherapy, biological agent, or investigational drug for SCLC.
* The patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* The patient is 18 years of age or older at the time informed consent is obtained.
* The patient must be accessible for study treatment and follow-up. Patients enrolled in this study must be treated at participating study centers for all 3 days of study drug administration in either treatment group.
* The patient has normal organ function.
* Women of childbearing potential must have a negative serum pregnancy test 72 hours prior to study enrollment. Women of childbearing potential and men with partners of childbearing potential must use a highly effective method of contraception throughout the entire study and up to 8 weeks after the last dose of any study drug (including obatoclax maintenance). Effective contraception or birth control is defined as those with a low failure rate (less than 1% per year) when used consistently and correctly.
* Women must not be breastfeeding.
* Written informed consent is obtained.
* Patients with asymptomatic brain metastases may be enrolled and if clinically indicated, may be treated with steroids to be tapered as tolerated by the patient. Patients with symptomatic brain metastases will be eligible for the study after they have received therapeutic whole brain irradiation (WBI), which must be completed at least 7 days before the day of first treatment with study drugs. Since these patients will also be treated with steroids it is recommended that steroids be tapered as clinically indicated and tolerated by the patient. The use of chronic, low-dose steroids is not contraindicated for these patients (or any other patients). Stereotactic radiation will be allowed for 1 to 3 brain metastatic lesions that meet appropriate criteria for that procedure; however, this must be discussed with the study monitor prior to consideration for enrollment into this study.
* The patient must be willing and able to comply with study restrictions and to remain at the study center for the required duration during the study period and willing to return to the study center for the follow-up evaluation as specified in this protocol.

Exclusion Criteria:

* The patient has had any prior systemic therapy for ES-SCLC other than radiation therapy or surgery.
* The patient has a history of prior malignancy with the exception of cervical intraepithelial neoplasia, basal cell or squamous cell carcinoma of the skin, or other localized malignancy that has undergone potentially curative therapy and is deemed by his or her treating physician to be at low risk for recurrence for 5 years.
* The patient has a history of hypersensitivity or allergic reactions attributed to components of the obatoclax mesylate formulation (ie, polysorbate 20 and polyethylene glycol [PEG] 300) or to carboplatin or etoposide.
* The patient currently has leptomeningeal disease or paraneoplastic syndromes.
* The patient has uncontrolled intercurrent illness including, but not limited to, symptomatic neurologic illness; active, uncontrolled systemic infection considered opportunistic, life-threatening, or clinically significant at the time of treatment; symptomatic congestive heart failure; unstable angina pectoris; clinically significant cardiac arrhythmia; significant pulmonary disease or hypoxia; or psychiatric illness that would limit compliance with study requirements.
* The patient is a pregnant or lactating woman. (Any women becoming pregnant during the study will be withdrawn from the study but will be monitored for safety.)
* The patient has a positive test result for hepatitis B surface antigen (HBsAg) or antibodies to hepatitis C virus (HCV Ab) or a known positive history of antibodies to human immunodeficiency virus (HIV) and is receiving combination antiretroviral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2016-05 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS): Time to Death | 24 months from last patient enrolled
  After 570 death events have been observed (Interim Analysis after 171 death events)or 24 months from last patient enrolled

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 24 months from last patient enrolled
  Randomization to Date of First Documented Disease Progression or Death for up to 24 months from last patient enrolled
Duration of Response | 24 months from last patient enrolled
  First Response to Disease Progression or Death up to 24 months from last patient enrolled
Objective Response Rate (Complete Response or Partial Response) | 37 months
Quality of Life | 37 months
  This is assessed with the European Organization for Research and Treatment of Cancer(EORTC)QLQ-C30 and EORTC QLQ-LC13 questionnaires